CLINICAL TRIAL: NCT02279875
Title: A Phase 2 Dose-ranging Trial to Evaluate the Bactericidal Activity, Safety, Tolerability and Pharmacokinetics of Linezolid in Adult Subjects With Newly Diagnosed Drug-Sensitive, Smear-Positive Pulmonary Tuberculosis.
Brief Title: A Phase 2 Trial to Evaluate the Efficacy and Safety of Linezolid in Tuberculosis Patients. (LIN-CL001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIN-CL001
Record Dates: First submitted 2014-10-28; First posted 2014-10-31 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Tuberculosis
Keywords: Tuberculosis; Drug-Sensitive Tuberculosis; Linezolid; HRZE (isoniazid, rifampicin, pyrazinamide, ethambutol); Pulmonary Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Linezolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Linezolid 300 mg once per day (Experimental): Half of a 600mg (scored) tablet
  Interventions: Drug: Linezolid
- Linezolid 300 mg twice per day (Experimental): Half of a 600mg (scored) tablet
  Interventions: Drug: Linezolid
- Linezolid 600 mg once per day (A) (Experimental): 600mg (scored) tablet
  Interventions: Drug: Linezolid
- Linezolid 600 mg once per day (B) (Experimental): 600mg (scored) tablet
  Interventions: Drug: Linezolid
- Linezolid 600 mg twice per day (Experimental): 600mg (scored) tablet
  Interventions: Drug: Linezolid
- Linezolid 1200 mg once per day (Experimental): Two 600mg (scored) tablets
  Interventions: Drug: Linezolid
- Linezolid 1200 mg 3 times per week (Experimental): Linezolid 1200 mg administered as a single oral dose three times per week (1200 mg: Day 1, 3, 5, 8, 10, and 12)
  Interventions: Drug: Linezolid
- HRZE once per day (Active Comparator): Treatment will be administered orally once daily for 14 days per the
  Subject's weight as follows:
  30-37 kg: 2 tablets;
  38-54 kg: 3 tablets;
  55-70 kg: 4 tablets;
  71 kg and over: 5 tablets.
  Interventions: Drug: HRZE (isoniazid rifampicin,pyrazinamide,ethambutol)

INTERVENTIONS:
Drug: Linezolid
  Arms: Linezolid 1200 mg 3 times per week; Linezolid 1200 mg once per day; Linezolid 300 mg once per day; Linezolid 300 mg twice per day; Linezolid 600 mg once per day (A); Linezolid 600 mg once per day (B); Linezolid 600 mg twice per day
Drug: HRZE (isoniazid rifampicin,pyrazinamide,ethambutol) — isoniazid (H) 75 mg plus rifampicin (R) 150 mg plus pyrazinamide (Z) 400 mg plus ethambutol (E) 275 mg
  Arms: HRZE once per day

SUMMARY:
The purpose of this study is to evaluate the mycobactericidal activity, safety, tolerability, and pharmacokinetics of 6 doses of linezolid: 300 mg once per day, 300 mg twice per day, 600 mg once per day, 600 mg twice per day and 1200 mg once per day administered orally for 14 consecutive days or 1200 mg administered three times per week for two weeks in adult subjects with newly diagnosed drug-sensitive, smear-positive pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

Subjects are required to meet all of the following inclusion criteria in order to be randomized.

1. Provide written, informed consent prior to all trial-related procedures.
2. Male or female, aged between 18 and 75 years inclusive.
3. Body weight (in light clothing and with no shoes) between 35 and 100 kg, inclusive.
4. Drug-sensitive pulmonary Tuberculosis (TB) determined by testing at the trial appointed laboratory: M.tb positive and rifampicin sensitive on molecular test (e.g. GeneXpert or Hain) and sputum smear-positive pulmonary TB on direct microscopy for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale).

   1. either newly diagnosed OR
   2. untreated for at least 3 years after cure from a previous episode (Subject can give a history of cure and previous treatment); AND
   3. Previous TB treatment must be discontinued as per exclusion criteria 17.
5. A chest X-Ray which in the opinion of the Investigator is consistent with TB.
6. Ability to produce an adequate volume of sputum as estimated from a screening Coached Spot Sputum Sample assessment (estimated 10 ml or more overnight production).
7. Be of non-childbearing potential or using effective methods of birth control, as defined below:

Non-childbearing potential:

1. Subject - not heterosexually active or practices sexual abstinence; OR
2. Female Subject/sexual partner - bilateral oophorectomy, bilateral tubal ligation and/or hysterectomy or has been postmenopausal with a history of no menses for at least 12 consecutive months; OR
3. Male Subject/sexual partner - vasectomised or has had a bilateral orchidectomy minimally three months prior to screening;

Effective birth control methods:

A double contraceptive method should be used as follows:

1. Double barrier method which can include any 2 of the following: a male condom, diaphragm, cervical cap, or female condom (male and female condoms should not be used together); OR
2. Barrier method (one of the above) combined with hormone-based contraceptives or an intra-uterine device for the female Subject/partner; AND
3. Are willing to continue practicing one of the above mentioned birth control methods throughout treatment and for 1 month (both male and female Subjects) after the last dose of study medication or discontinuation from study medication in case of premature discontinuation.

Exclusion Criteria:

Subjects will be excluded from participation if they meet any of the following criteria.

Medical Criteria

1. Evidence of clinically significant (as judged by the Investigator), metabolic, gastrointestinal, cardiovascular, musculoskeletal, ophthalmological, pulmonary, neurological, psychiatric or endocrine diseases, malignancy, or other abnormalities (other than the indication being studied) including malaria.

   A rapid test for malaria may be carried out if indicated.
2. Poor general condition where any delay in treatment cannot be tolerated per discretion of the Investigator.
3. Clinically significant evidence of extrathoracic TB (e.g. miliary TB, abdominal TB, urogenital TB, osteoarthritic TB, TB meningitis), as judged by the Investigator.
4. History of allergy or hypersensitivity to any of the study Investigational Medicinal Products or related substances.
5. Known or suspected current alcohol and/or drug abuse (positive urine drug screen) or history thereof within the past 2 years that is, in the opinion of the Investigator, sufficient to compromise the safety and/or cooperation of the Subject.
6. A history of seizures or risk factors for seizures.
7. For HIV infected Subjects:

   1. having a CD4+ count <250 cells/μL;
   2. with an AIDS-defining opportunistic infection or malignancies (except pulmonary TB);
   3. OR having received antiretroviral therapy medication within the last 90 days
   4. OR having received oral or intravenous antifungal medication within the last 90 days.
8. Having participated in other clinical study/ies with investigational agent/s within 8 weeks prior to trial start.
9. Significant cardiac arrhythmia requiring medication or QT interval on ECG >500msec on screening ECG.
10. Subjects with uncontrolled hypertension, pheochromocytoma, thyrotoxicosis
11. Females who are pregnant or breast-feeding, or planning to conceive a child during the study or within 1 month of cessation of treatment
12. Diabetes Mellitus

    Specific Treatments
13. Previously received treatment with linezolid.
14. Known allergy or intolerance to linezolid.
15. Concomitant use of monoamine oxidase inhibitors (MAOIs) or prior use within 1 month of screening.
16. Concomitant use of serotonergic agents including SSRI/SNRI antidepressants or prior use within 3 days of screening should be avoided if possible as subjects on these agents and linezolid are at risk for serotonin syndrome.
17. Treatment with any drug active against M.tb within 3 months prior to Day 1 (including but not limited to isoniazid, ethambutol, amikacin, bedaquiline, clofazimine, cycloserine, fluoroquinolones, rifabutin, rifampicin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, pyrazinamide, thioacetazone, capreomycin, thioamides, metronidazole).

    Based on Laboratory Abnormalities:
18. Subjects with the following toxicities at screening as defined by the enhanced Division of Microbiology and Infectious Disease (DMID) adult toxicity table (November 2007):

    1. creatinine grade 2 or greater [>1.5 x Upper Limit of Normal (ULN)];
    2. hemoglobin level of <8.0 gm/dL;
    3. platelet count <80,000/mm3;
    4. absolute neutrophil count <1000/mm3
    5. serum potassium, serum magnesium and calcium (corrected for albumin) levels less than the lower limit of normal for the laboratory;
    6. aspartate aminotransferase (AST) grade 3 or greater (≥3.0 x ULN) to be excluded;
    7. alanine aminotransferase (ALT) grade 3 or greater (≥3.0 x ULN) to be excluded;
    8. alkaline phosphatase (ALP) grade 4 (>8.0 x ULN) to be excluded, grade 3 (≥3.0 - 8.0 x ULN) must be discussed with and approved by the Sponsor Medical Monitor;
    9. total bilirubin grade 3 or greater (≥2.0 x ULN, or ≥1.50 x ULN when accompanied by any increase in other liver function test) to be excluded, grade 2 (≥1.50 x ULN, or ≥1.25 x ULN when accompanied by any increase in other liver function test) must be discussed with and approved by the Sponsor Medical Monitor;

Any laboratory value which excludes the Subject may be repeated to confirm eligibility.

All inclusion and no exclusion criteria must be met. If no single variable/value is outside of the ranges of acceptability, but when multiple values are close to the limits and/or whenever the Investigator has reason to suspect that there might be a health problem (other than TB), enrollment should only be considered after discussing the case with the sponsor medical monitor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Bactericidal Activity (Time to Positivity) Days 0 - 14 [BA(TTP)] | Days -2, -1, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
  [BA(TTP)] will be determined by the rate of change in time to sputum culture positivity (TTP) over 14 days of treatment in the Mycobacterial Growth Indicator Tube system, represented by the model-fitted log(TTP) results as calculated by the regression of the observed log(TTP) results over time.

SECONDARY OUTCOMES:
The Bactericidal Activity (Time to Positivity) Days 0 - 2 [BA(TTP)](0-2), and Bactericidal Activity (Time to Positivity) Days 7 - 14 [BA(TTP)](7-14) | Day -2, -1, 1, 2, 7, 8, 9, 10, 11, 12, 13, 14
  [BA(TTP)] will be determined by the rate of change in TTP represented by the model-fitted log(TTP) as calculated by the regression of the observed log(CFU) counts over time.
The Bactericidal Activity Colony Forming Unit (BACFU)(0-14), BACFU(0-2) and BACFU(7-14) | Day 1, 2, 3, 4, 5, 6, 7, 8, 8, 9, 10, 11, 12, 13, 14
  [BACFU] will be determined by the rate of change in colony forming unit (CFU) counts, over 14 days of treatment represented by the model-fitted log(CFU) counts as calculated by the regression of the observed log (CFU) counts over time.
Incidence of Treatment Emergent Adverse Events (TEAEs) presented by severity (DMID Grade), relatedness, and seriousness, leading to early withdrawal and leading to death. | Screening (-9 to -3, -2, -1), Day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, and Follow-Up (Day 21)
Pharmacokinetic parameters for subjects (except in the HRZE treatment arm): Cmax, T1/2, AUC 0 - 12 | Day 12 (pre-dose, 0.5, 1, 2, 4, 8, 12 and 24 hours post-dose) for 1200 3X per week, Day 14 (pre-dose, 0.5, 1, 2, 4, 8, 12, and 24 hours post-dose) for 600 mg QD (B), and Day 14 (pre-dose, 0.5, 1, 2, 4, 8, and 12 hours post-dose) for other arms
  Cmax: Maximum observed plasma drug concentration. T1/2: Half-life of elimination of the profile. AUC0-12: Area under the concentration time (t) curve from zero to 12 hours. Before calculation of AUC0-12, the 12 hour post-dose concentration will be interpolated using T1/2, if not available
Time over minimum inhibitory concentration (MIC) will be calculated for each subject in the linezolid arms individually and for each of the linezolid arms as a group, based on the MIC determined at baseline. | Baseline (Day -2 to -1), Day 12 (1200 mg three times per week), Day 14 (all other experimental arms)
Time over concentration that inhibits 50% of mitochondrial protein synthesis (MPS IC50) | Day 12 (1200 mg three times per week), Day 14 (all other experimental arms)
  calculated for each subject in the linezolid arms individually and for each of the linezolid arms as a group, based on the established MPS IC50 for linezolid (8.0 ug/ml).
Correlation between AUC0-12 and AUC0-inf, Cmax and time over minimum inhibitory concentration and BA (0-2, 0-14 and 7-14) will be determined using both time to positivity and colony forming unit results, for all subjects combined. | Days -2, -1, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14

CONTACTS AND LOCATIONS:
Overall Officials: Christo van Niekerk, Study Director — Global Alliance for TB Drug Development; Adreas Diacon, Principal Investigator — Task Clinical Research Centre; Rod Dawson, Principal Investigator — University of Cape Town Lung Institute (Pty) Ltd
Locations (2):
- South Africa (2):
  - TASK Clinical Research Centre, Bellville, Cape Town
  - University of Cape Town Lung Institute (Pty) Ltd, Mowbray, Cape Town

REFERENCES:
- [Derived] Simeon S, Garcia-Cremades M, Savic R, Solans BP. Pharmacokinetic-pharmacodynamic modeling of tuberculosis time to positivity and colony-forming unit to assess the response to dose-ranging linezolid. Antimicrob Agents Chemother. 2024 Aug 7;68(8):e0019024. doi: 10.1128/aac.00190-24. Epub 2024 Jul 17. PMID 39016594
- [Derived] Diacon AH, De Jager VR, Dawson R, Narunsky K, Vanker N, Burger DA, Everitt D, Pappas F, Nedelman J, Mendel CM. Fourteen-Day Bactericidal Activity, Safety, and Pharmacokinetics of Linezolid in Adults with Drug-Sensitive Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e02012-19. doi: 10.1128/AAC.02012-19. Print 2020 Mar 24. PMID 31988102
- See also: TB Alliance Website — http://www.tballiance.org